CLINICAL TRIAL: NCT02427685
Title: Dysfunctional Hemoglobin
Brief Title: Dysfunctional Hemoglobin CO-ox
Status: Completed | Type: Observational
Sponsor: Nonin Medical, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: QATP2687
Record Dates: First submitted 2015-04-20; First posted 2015-04-28 (Estimated); Last update posted 2015-06-17 (Estimated); Status verified 2015-04

CONDITIONS: Elevated Levels of Carboxyhemoglobin

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Pulse Co-Ox — Comparison of pulse co-oximeter to blood gas analyzer.

SUMMARY:
The study verifies accuracy of a new pulse co-oximeter in the presence of elevated carboxyhemoglobin levels.

ELIGIBILITY:
Inclusion Criteria:

* The subject is male or female.
* The subject is of any racial or ethnic group.
* The subject is between 18 years and 45 years of age.
* The subject does not have significant medical problems.
* The subject is willing to provide written informed consent and is willing and able to comply with study procedures.

Exclusion Criteria:

* Has a BMI greater than 31
* Has had any relevant injury at the sensor location site
* Has deformities or abnormalities that may prevent proper application of the device under test.
* Has a known respiratory condition.
* Is currently a smoker.
* Has a known heart or cardiovascular condition.
* Is currently pregnant.
* Is female and actively trying to get pregnant.
* Has a clotting disorder.
* Has Raynaud's Disease.
* Is known to have a hemoglobinopathy such as (anemia, bilirubinemia, sickle-cell anemia, inherited or congenital methemoglobinemia).
* The subject has a COHb greater than 3% or MetHb greater than 2%.
* Has taken blood thinners or medication with aspirin within the last 24 hours.
* Has unacceptable collateral circulation from the ulnar artery.
* Has donated more than 300 mL of blood within one month prior to start of study.
* Is unwilling or unable to provide written informed consent to participate in the study.
* Is unwilling or unable to comply with the study procedures for the primary objectives.
* Has another health condition which in the opinion of the principal investigator makes him/her unsuitable for testing.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adult volunteers
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2015-04; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Carboxyhemoglobin over the range of 0-15 percent as assessed by co-oximetry. | 3 hours

SECONDARY OUTCOMES:
Oxygen saturation accuracy in conditions of elevated carboxyhemoglobin. | 3 hours

CONTACTS AND LOCATIONS:
Overall Officials: Phillip E Bickler, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States